CLINICAL TRIAL: NCT00395057
Title: A Study Using Intravitreal Injections of a Small Interfering RNA in Patients With Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to company decision (non-safety related).
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 211745-001
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Results first posted 2011-12-13 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Choroid Neovascularization; Age-Related Macular Degeneration
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (4):
- AGN 211745 Solution 1000 ug (Experimental): AGN 211745 Solution 1000 ug
  Interventions: Drug: AGN 211745
- AGN 211745 Solution 300 ug (Experimental): AGN 211745 Solution 300 ug
  Interventions: Drug: AGN 211745
- AGN 211745 Solution 100 ug (Experimental): AGN 211745 Solution 100 ug
  Interventions: Drug: AGN 211745
- Ranibizumab 500 ug (Active Comparator): Ranibizumab 500 ug
  Interventions: Drug: Ranibizumab 500µg

INTERVENTIONS:
Drug: AGN 211745 — AGN 211745 Solution 1000µg injection at Day 1, Month 1, Month 2
  Other Names: Sirna-027
  Arms: AGN 211745 Solution 1000 ug
Drug: AGN 211745 — AGN 211745 Solution 300µg injections, Day 1, Month 1, Month 2
  Other Names: Sirna-027
  Arms: AGN 211745 Solution 300 ug
Drug: AGN 211745 — AGN 211745 Solution 100µg injections, Day 1, Month 1, Month 2
  Other Names: Sirna-027
  Arms: AGN 211745 Solution 100 ug
Drug: Ranibizumab 500µg — Ranibizumab 500µg injections at Day 1, Month 1, Month 2
  Other Names: Lucentis®
  Arms: Ranibizumab 500 ug

SUMMARY:
This is a 24-month study to evaluate multiple doses of AGN211745 (previously known as Sirna-027) in treatment of subfoveal choroidal neovascularization associated with age-related macular degeneration

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older with "wet" AMD as determined by an ophthalmologist
* decrease in visual acuity (20/40 to 20/640) in at least one eye

Exclusion Criteria:

* Uncontrolled systemic disease
* History of heart attack or stroke within one year of study entry
* Symptomatic coronary artery disease
* Cataracts that interfere with vision

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2007-01; Primary Completion 2008-10 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (3):
- Houston, Texas, United States
- Sydney, New South Wales, Australia
- Makati, Philippines

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AGN 211745 Solution 1000 ug | AGN 211745 Solution 300 ug | AGN 211745 Solution 100 ug | Ranibizumab 500 ug
Started | 34 | 35 | 35 | 34
Completed | 2 | 1 | 2 | 1
Not Completed | 32 | 34 | 33 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN 211745 Solution 1000 ug | AGN 211745 Solution 300 ug | AGN 211745 Solution 100 ug | Ranibizumab 500 ug | Total
Number analyzed (Participants) | 34 | 35 | 35 | 34 | 138
Age, Customized [Number; unit: participants]
  Between 45 and 65 years | 2 | 5 | 5 | 4 | 16
  >=65 years | 32 | 30 | 30 | 30 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 24 | 14 | 76
  Male | 15 | 16 | 11 | 20 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Improvement in Best Corrected Visual Acuity (BCVA) of 15 or More Letters at Month 3
Description: Percentage of patients with improvement in BCVA of 15 or more letters at Month 3. BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Time Frame: Month 3
Population: Intent-To-Treat (ITT). The ITT population included all patients who started the study (randomized).
Measure: Number; unit: Percentage of Patients
Arm/Group | AGN 211745 Solution 1000 ug | AGN 211745 Solution 300 ug | AGN 211745 Solution 100 ug | Ranibizumab 500 ug
Number analyzed (Participants) | 34 | 35 | 35 | 34
Percentage of Patients | 5.9 | 2.9 | 0 | 17.6

2. Secondary Outcome: Lesion Size as Assessed by Fluorescein Angiography (FA) and Photography at Month 3
Description: Lesion size as assessed by FA and photography at month 3. FA is a technique for examining the circulation of the retina (and detecting any leakage) using a dye-tracing method. Photographs are taken with a specialized low-power microscope with an attached camera designed to photograph the interior of the eye, including the retina and optic disc.
Time Frame: Month 3
Population: Intent-To-Treat. The ITT population included all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Millimeters squared (mm^2)
Arm/Group | AGN 211745 Solution 1000 ug | AGN 211745 Solution 300 ug | AGN 211745 Solution 100 ug | Ranibizumab 500 ug
Number analyzed (Participants) | 34 | 35 | 35 | 34
Millimeters squared (mm^2) | 6.17 (4.339) | 4.29 (3.264) | 6.54 (6.102) | 3.89 (3.396)

3. Secondary Outcome: Foveal Thickness as Assessed by Optical Coherence Tomography (OCT) at Month 3
Description: Foveal thickness as assessed by OCT at month 3. The fovea is a part of the eye, located in the center of the macula region of the retina. OCT is a laser-based, noninvasive, diagnostic system providing high-resolution, three-dimensional images of the retina. The fovea is responsible for sharp central vision, which is necessary for reading or any activity where visual detail is of primary importance. Normal foveal thickness ranges from 175 to 250 microns. A foveal thickness greater than 250 microns represents worsening vision.
Time Frame: Month 3
Population: Intent-To-Treat (ITT). The ITT population included all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | AGN 211745 Solution 1000 ug | AGN 211745 Solution 300 ug | AGN 211745 Solution 100 ug | Ranibizumab 500 ug
Number analyzed (Participants) | 34 | 35 | 35 | 34
Microns | 484.6 (142.21) | 413.2 (103.59) | 437.1 (125.46) | 269.8 (76.72)

4. Secondary Outcome: Visual Functioning Questionnaire (VFQ) at Month 3
Description: Visual Functioning Questionnaire (VFQ) at Month 3. The VFQ includes 25 questions which assess visual impairment on functioning and specific aspects of health-related quality of life. Study terminated; data for this outcome measure were not analyzed.
Time Frame: Month 3
Population: Intent-To-Treat (ITT). The ITT population included all patients who started the study (randomized). Data for this outcome measure were not analyzed as the study was terminated early.
Arm/Group | AGN 211745 Solution 1000 ug | AGN 211745 Solution 300 ug | AGN 211745 Solution 100 ug | Ranibizumab 500 ug
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Time to Treatment With Standard of Care at Month 6
Description: Time to treatment with standard-of-care at month 6, defined as the number of days before the use of rescue therapy occurred.
Time Frame: Month 6
Population: Intent-To-Treat (ITT). The ITT population included all patients who started the study (randomized).
Measure: Median (95% Confidence Interval); unit: Number of Days
Arm/Group | AGN 211745 Solution 1000 ug | AGN 211745 Solution 300 ug | AGN 211745 Solution 100 ug | Ranibizumab 500 ug
Number analyzed (Participants) | 34 | 35 | 35 | 34
Number of Days | 91.0 [86.00 to 102.0] | 91.5 [90.00 to 119.0] | 92.0 [91.00 to 112.0] | 130.5 [96.00 to 161.0]

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for SAEs and AEs and is the total number of patients that were randomized AND treated.
Arm/Group | AGN 211745 Solution 1000 ug | AGN 211745 Solution 300 ug | AGN 211745 Solution 100 ug | Ranibizumab 500 ug
Serious Adverse Events (participants affected / at risk) | 4/34 | 3/35 | 3/35 | 9/34
Other Adverse Events (participants affected / at risk) | 29/34 | 26/35 | 28/35 | 24/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGN 211745 Solution 1000 ug (N=34) | AGN 211745 Solution 300 ug (N=35) | AGN 211745 Solution 100 ug (N=35) | Ranibizumab 500 ug (N=34)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Biliary tract disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster ophthalmic (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN 211745 Solution 1000 ug (N=34) | AGN 211745 Solution 300 ug (N=35) | AGN 211745 Solution 100 ug (N=35) | Ranibizumab 500 ug (N=34)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 2
Conjunctival haemorrhage (Eye disorders) | 10 | 9 | 12 | 5
Retinal haemorrhage (Eye disorders) | 5 | 2 | 2 | 3
Eye Pain (Eye disorders) | 3 | 9 | 5 | 1
Anterior chamber cell (Eye disorders) | 3 | 2 | 1 | 1
Conjunctival oedema (Eye disorders) | 3 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 2 | 4 | 2 | 3
Vitreous floaters (Eye disorders) | 2 | 2 | 5 | 0
Conjunctival hyperaemia (Eye disorders) | 2 | 2 | 4 | 2
Detachment of retinal pigment (Eye disorders) | 2 | 5 | 1 | 2
Ocular discomfort (Eye disorders) | 2 | 0 | 0 | 1
Retinal neovascularization (Eye disorders) | 2 | 0 | 0 | 1
Retinal exudates (Eye disorders) | 2 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 1 | 5 | 0 | 1
Anterior chamber flare (Eye disorders) | 1 | 2 | 0 | 1
Retinal oedema (Eye disorders) | 1 | 1 | 2 | 3
Macular degeneration (Eye disorders) | 1 | 0 | 1 | 2
Vitreous detachment (Eye disorders) | 0 | 4 | 1 | 1
Vision blurred (Eye disorders) | 0 | 3 | 2 | 1
Eye irritation (Eye disorders) | 0 | 2 | 3 | 1
Blepharitis (Eye disorders) | 0 | 2 | 1 | 1
Eye discharge (Eye disorders) | 0 | 2 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 1 | 2 | 1
Retinal pigment epitheliopathy (Eye disorders) | 0 | 0 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 2 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 3 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to a company decision (non-safety related). Because the study was terminated early, data for certain outcome measures (ie, "Visual Functioning Questionnaire [VFQ] at Month 3") were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo